CLINICAL TRIAL: NCT01563835
Title: Analgesia for 2nd Trimester Termination of Pregnancy: a Randomized Controlled Trial of Intravenous Versus Epidural Patient Controlled Analgesia
Brief Title: Analgesia for 2nd Trimester Termination of Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: Termination of pregnancy; Epidural; IV PCA
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural (PCEA) (Active Comparator): bupivacaine, fentanyl
  Interventions: Drug: bupivacaine, fentanyl
- IV PCA (Active Comparator): Intravenous fentanyl patient controlled analgesia
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: bupivacaine, fentanyl — 10mL of 0.125% of bupivacaine plus 50 mcg fentanyl, injected through an epidural catheter.
  Other Names: bupivacaine: Marcaine; fentanyl: fentanyl citrate
  Arms: Epidural (PCEA)
Drug: fentanyl — fentanyl IV PCA with boluses 25-50 mcg, 3-6 minute lockout.
  Other Names: fentanyl citrate
  Arms: IV PCA

SUMMARY:
There has been very little investigation into the management of pain from 2nd trimester termination of pregnancy or unexpected fetal loss. The standard of practice in North America is usually intravenous patient controlled analgesia (IV PCA), using a narcotic wuch as fentanyl. The goal of this study is to compare the quality of recovery after termination of pregnancy using fentanyl IV PCA or patient controlled epidural analgesia (PCEA), a standard of care for live births. The study will be conducted as a randomized controlled trial.

DETAILED DESCRIPTION:
Epidural analgesia is known to provide superior analgesia for labour with minimal maternal and fetal side effects. This mode of analgesia is not usually offered to patients who require termination of their pregnancies or who suffer unexpected fetal losses, although they go through labour and delivery with likely more difficult psychological circumstances.

We plan to compare patient controlled epidural analgesia (PCEA) with intravenous patient controlled analgesia (IV PCA), for 2nd trimester terminations of pregnancy. We hypothesize that PCEA provides better quality of recovery than IV PCA. The previously validated Quality of Recovery - 40 questionnaire will be used to measure a patient's quality of recovery. The results of this study will determine the optimal method of pain relief for late termination of pregnancy or fetal loss.

ELIGIBILITY:
Inclusion Criteria:

* interruption of pregnancy between 12 and 23 6/7 weeks

Exclusion Criteria:

* documented allergy to fentanyl or bupivacaine
* coagulopathy
* drug or narcotic abuse
* contraindication to neuraxial analgesia
* inability to comply with IVPCA or PCEA
* inability to complete the QoR-40 questionnaire
* TOP due to maternal problems

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery - 40 score on discharge | up to 5 days
  The primary outcome of this study will be the difference between IV PCA and PCEA groups in aggregate score of Quality of Recovery - 40 on discharge from hospital.

SECONDARY OUTCOMES:
Duration of procedure | 24 hours
  Duration of procedure from induction to abortion in hours
Pain score | 24 hours
  Visual analog pain score every 30 minutes during procedure
Narcotic-related complications | 24 hours
  Incidence of: nausea/vomiting, pruritis, sedation, respiratory depression.
Epidural-related complications | 24 hours
  Incidence of: hypotension, dural puncture, local anesthetic toxicity, neurological complications.
Surgical intervention | 24 hours
  Incidence of surgical intervention and any anesthetic required for intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada